CLINICAL TRIAL: NCT05033301
Title: Virtualizing Survivorship: Implementing a More Timely and Comprehensive Model of Follow-up Care: Effectiveness Evaluation Phase
Brief Title: Evaluating the Effectiveness of the Nurse Ned Clinic
Acronym: NurseNed
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Trillium Health Partners (Other); Niagara Health System (Other); Alberta Health services (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-5188
Record Dates: First submitted 2021-08-21; First posted 2021-09-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Digital Health; Nurse-led Care Model; Survivorship Care
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specialist-led Ned Clinic (No Intervention): Participants enrolled in specialist-led version of the Ned Virtual Clinic will be prompted to complete their PROs (EPIC-26 survey) and PSA/testosterone lab tests in accordance to their pre-specified follow-up surveillance protocol determined by the specialist for one year.
- Nurse-led Ned Clinic (Experimental): Participants enrolled in the nurse-led version of the Ned Virtual Clinic will be prompted to complete their PROs (EPIC-26 survey) and PSA/testosterone lab tests in accordance to their pre-specified follow-up surveillance protocol determined by the specialist. In addition, men will be asked to complete another set of PROs that will be monitored by a trained oncology nurse, in between their specialist visits.
  Interventions: Device: Nurse Ned Clinic

INTERVENTIONS:
Device: Nurse Ned Clinic — Participants enrolled in the Nurse-led Ned Clinic will receive virtual PCa survivorship follow-up care from both their specialist and an oncology nurse for one year.
  Arms: Nurse-led Ned Clinic

SUMMARY:
The purpose of this non-randomized control trial is to evaluate the effectiveness of a virtual nurse-led survivorship clinic for prostate cancer (PCa) survivors. Through this trial, investigators will compare pre-determined survivorship outcomes of men receiving care via traditional specialist-led PCa virtual care model (Specialist Ned) to those receiving care via the newly-proposed nurse-led PCa virtual care model (Nurse Ned). In total, it is anticipated that a maximum of 600 men (300 in control arm; 300 in intervention arm) across five clinical sites (3 in Ontario; 1 in Alberta; and 1 in Nova Scotia) will be enrolled into this trial and will be followed for 12 months.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common cancer among Canadian men, with over 25,000 diagnosed yearly. While advances in treatment and care, including the PSA (prostate-specific antigen) test have resulted in more men entering survivorship and living longer, many continue to experience undesirable symptoms, side effects and psychosocial concerns. The current healthcare system is not optimized to deliver survivorship care at scale and struggles to support the increasing number of survivors across the cancer care continuum. Increasing patient loads in specialty clinics result in brief and infrequent follow-up visits, leaving patients without the opportunity to ask questions and fully understand their health status, all the while tasking providers with making quick and effective treatment decisions with minimal patient information or interaction.

In order to address this increasing need for improved care delivery, investigators have developed the Ned ("No Evidence of Disease") PCa survivorship platform, which allows patients to access clinical information (i.e. lab results), virtually complete patient reported outcomes (PROs) on their quality of life, and complete virtual visits with their specialist. Despite the promise and potential of Ned, ongoing evaluation of this platform shows specialists often lacked the availability and flexibility to consistently review ePROs and lab results prior to a study visit. In response, researchers aim to expand the current Ned platform to design, develop and implement a digitally mediated nurse-led survivorship care model that can address the growing needs of prostate cancer survivors and healthcare providers at scale.

In this trial, investigators aim to evaluate the effectiveness of a nurse-led survivorship care model by comparing the clinical outcomes of patients enrolled in the Specialist Ned Clinic (control) for their PCa follow-up care and those that will be enrolled into the Nurse Ned Clinic (intervention) a year later. Participants will be enrolled in the study for one year, and will be asked to complete standardized questionnaires related to their PCa follow-up care at the start of the study, 6-months into using their respective Ned Clinic and at study completion.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Completed curative-intent treatment
3. Receiving PCa survivorship care at University Health Network (UHN), Trillium Health Partners (THP), Niagara Health System (NHS), Prostate Cancer Centre - Calgary (PCCC), or Queen Elizabeth II Health Sciences Centre (QEII HSC)-affiliated hospital
4. Low risk of recurrence as determined by their treatment specialist
5. Adequate English ability (or a caregiver willing to provide translation) to complete study activities as determined by research assistant
6. Have an email address (or be able to use the email address of a caregiver)

Exclusion Criteria:

Patients with metastatic PCa are not eligible to participate in this research.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in unmet needs | Measured at Baseline, 6 months, 1 year
  Assessed by Cancer Survivors' Unmet Needs (CaSUN) questionnaire. The questionnaire is a 42-item instrument that captures the current needs of a cancer survivor, such as medical care, quality of life, emotional and relationship needs and their current view of life.

SECONDARY OUTCOMES:
Changes to Participant's Health Status | Measured at Baseline, 6 months, 1 year
  Assessed by the EQ5D-5L questionnaire. This questionnaire contains 6 questions which assess the patient's health status by understanding how they feel about their mobility, self-care, usual activities, pain/discomfort and levels of anxiety or depression.
Changes in Prostate Cancer health related quality of life | Measured at Baseline, 6 months, 1 year
  Assessed by the Expanded Prostate Cancer Index Composite Short Form (EPIC-26). The questionnaire is a 13-item instrument that captures the side effects and symptoms that might affect the quality of life in patients with prostate cancer patients.
Changes in overall health related quality of life | Measured at Baseline, 6 months, 1 year
  Assessed by the Functional Assessment of Cancer Therapy for Prostate Cancer patients (FACT-P). This questionnaire is a 39-item instrument that assesses the quality of health-related well-being for patients with prostate cancer.
Changes in Psychological Wellbeing | Measured at Baseline, 6 months, 1 year
  Assessed by the General Health Questionnaire (GHQ-12). This questionnaire contains 12-questions that ask prostate cancer patients how they have been feeling in the past weeks.
Changes in willingness to self-manage | Measured at Baseline and 1 year
  Assessed by the Patient Activation Measure Questionnaire (PAM-13). This questionnaire is a 13-item instrument that quantifies a patient's readiness to engage in their own self-management.
Changes to satisfaction with care | Measured at Baseline and 1 year
  Assessed by the Care Satisfaction Questionnaire. This questionnaire is an 11-item instrument used to quantify experience and acceptability of follow-up care.
Changes in health behaviours | Measured at Baseline and 1 year
  Assessed by the Health Behaviour Questionnaire. This questionnaire is used to determine participant health practices (e.g. smoking, fitness, alcohol consumption).

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network (Princess Margaret Hospital), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Findings from the study will be published and shared through open-accessed peer review journals and scientific conferences within the digital health and cancer respective fields. Results will be shared in aggregate.